Title: Brain Functioning and Decision-Making

NCT #: NCT03974282

Document date: 06/05/2019

Document Type: Informed Consent

# RESEARCH SUBJECT INFORMATION AND CONSENT FORM

**TITLE: Brain Functioning and Decision-Making** 

VCU IRB NO.: HM20015724

**INVESTIGATOR: Dr. David Chester** 

## **ABOUT THIS CONSENT FORM**

You are being invited to participate in a research study. It is important that you carefully think about whether being in this study is right for you and your situation.

This consent form is meant to assist you in thinking about whether or not you want to be in this study. Please ask the study staff to explain any information in this consent document that is not clear to you.

Your participation is voluntary. You may decide not to participate in this study. If you do participate, you may withdraw from the study at any time. Your decision not to take part or to withdraw will involve no penalty or loss of benefits to which you are otherwise entitled.

### PURPOSE OF THE STUDY

This study is about how brain function and structure is different between two universities. Your participation in this project will contribute to a better understanding of how universities affect the brain. This study will be completed in one, 3-hour laboratory visit today.

You are being invited to take part in this research study because you are 18 years old or older, meet comfort and safety criteria for an MRI environment, and are currently enrolled in a PSYC 101 course at VCU.

# **DESCRIPTION OF THE STUDY AND YOUR INVOLVEMENT**

If you decide to be in this research study, you will be asked to sign this consent form after you have had all your questions answered and understand what will happen to you.

In this study you will be asked to:

- 1. Complete an MRI safety screening form.
- 2. Practice the computer tasks that you will complete in the MRI scanner.
- 3. Enter the MRI scanner and complete a series of computer tasks while undergoing brain scans that measure the structure and functioning of your brain\*.
- 4. Complete a battery of questionnaires that will ask you about your personality.

Approved by the VCU IRB on 6/5/2019

\*MRI scans are a very common and safe form of brain imaging that use magnetic waves to record images of your body. While you lay inside of a large MRI machine, which looks like a large tube, we will pass magnetic waves through your head which can measure the structure and function of your brain. These procedures are very safe (for more information see the Risks and Discomforts section below).

Significant new findings developed during the course of the research which may relate to your willingness to continue participation will be provided to you. Approximately 100 people will participate in this study.

## **RISKS AND DISCOMFORTS**

To the best of our knowledge, the things you will be doing have no more risk of harm than you would experience in everyday life. You may find some questions we ask you (or some procedures we ask you to do) to be upsetting or stressful. You do not have to answer any questions that you do not want to, and you may leave the study at any time. If you become upset, the study staff will give you names of counselors to contact so you can get help in dealing with these issues.

Some procedures in this study may involve loud noises that may be uncomfortable or unpleasant, but which should not be physically harmful.

Participation in research might involve some loss of privacy. There is a small risk that someone outside the research study could see and misuse information about you.

The risks and discomforts of participating in the MRI study are outlined in the table below. Most of the risks are not serious, though there is a chance that we could find a serious abnormality in the structure of your brain. If an abnormality is found, and is indicative of a serious condition, the Principal Investigator (Chester) will contact you. A medical professional will be available to consult with you on how to proceed with this issue. It is important to note that the brain scans conducted in this study are NOT of clinical/diagnostic quality. As such, a scan from our study cannot be used to make a conclusive, medical diagnosis and a scan from this study that does not reveal any abnormalities should NOT prevent you from seeking medical testing if you are exhibiting symptoms of a suspected neurological issue. If an irregularity in your brain is found, the evaluation for this abnormality could lead to significant anxiety, costs and risks not included in this research study. Some abnormalities could affect your insurability or employability.

In addition to the risks below, you may experience a previously unknown risk or side effect:

| Possible | How often | How | Can it be corrected? |
|-----------|-----------|------------|----------------------|
| Risk/Side | has it | serious is | |

| Effect | occurred? | it? | |
|---|---|---|---|
| Claustrophobia | It | Can be | Yes, participant is removed |
| | occasionally | treated | from the magnet |
| | occurs | | |
| Dizziness | It | Not serious | Yes, change body positions |
| | occasionally | | slowly within the magnetic |
| | occurs | | field |
| Loud noise | It is expected | Not serious | Yes, participants wear ear |
| | to occur | | protection |
| Detection of a | It rarely | May be | Participant is told to contact |
| brain | occurs | serious | their primary care physician |
| abnormality | | | |

#### **BENEFITS TO YOU AND OTHERS**

You may not get any direct benefit from this study, but, the information we learn from people in this study may help us better understand human biology and behavior. In general, we do not have any plans to share your individual research results with you, aside from the sharing of any abnormalities in the MRI, as discussed above.

### COSTS

There are no costs for participating in this study other than the time you will spend completing the study.

### **PAYMENT FOR PARTICIPATION**

You will a thumbdrive with images of your brain. If you are currently enrolled in PSYC 101, you will receive 3.0 credit hours towards your PSYC 101 research requirement. If you are not currently enrolled in PSYC 101, you will receive \$40.

#### **ALTERNATIVES**

If you do not wish to complete this study, you can sign-up for other studies. If you are currently enrolled in PSYC 101, you can check your PSYC 101 syllabus for alternative means to complete your research requirement.

#### CONFIDENTIALITY

Potentially identifiable information about you will consist of your responses to a series of questionnaires, your responses to the computer tasks you perform in the MRI scanner, and images of your head and brain. Data is being collected only for research purposes.

All the other data listed above will be identified by ID numbers, not names, and stored on password-protected computers in a locked research area. All personal identifying information will be kept in password protected files and these files will be deleted immediately once the study is completed. Other records such as consent forms and data consent forms will be kept in a locked file cabinet for 5 years after the study ends and will be destroyed at that time. Your de-identified

data files will be kept indefinitely. Access to all data will be limited to study personnel.

What we find from this study may be presented at meetings or published in papers, but any of your identifying information will not ever be used in these presentations or papers. Your de-identified data from this study will be publicly-shared on the Open Science Framework (https://osf.io/), which is a website that allows others to view our data for the sake of scientific transparency. Your individual MRI images will never be shared outside of our approved research personnel, though aggregated MRI images that represent multiple participants from our study (and cannot be used to identify any one individual) will be publicly-shared on NeuroVault (https://neurovault.org/), which is a website that allows others to view our data for the sake of scientific transparency.

In the future, identifiers might be removed from the information you provide in this study, and after that removal, the information could be used for other research studies by this study team or another researcher without asking you for additional consent.

### **VOLUNTARY PARTICIPATION AND WITHDRAWAL**

Your participation in this study is voluntary, and there are no penalties for choosing not to participate or for withdrawing. If you would like to withdraw your data you can do so by contacting the Principal Investigator.

Your participation in this study may be stopped at any time by the study staff without your consent. The reasons might include:

- the study staff thinks it necessary for your health or safety;
- you have not followed study instructions
- administrative reasons require your withdrawal.

### **QUESTIONS**

If you have any questions, complaints, or concerns about your participation in this research, contact:

Dr. David Chester dschester@vcu.edu 804-828-7624

The researcher named above is the best person to call for questions about your participation in this study.

If you have any general questions about your rights as a participant in this or any other research, you may contact:

Office of Research Virginia Commonwealth University This Box for IRB Office Use Only – Do Not Delete or Revise Template Rev Date: 12-10-15

> 800 East Leigh Street, Suite 3000 Box 980568 Richmond, VA 23298 Telephone: (804) 827-2157

Contact this number to ask general questions, to obtain information or offer input, and to express concerns or complaints about research. You may also call this number if you cannot reach the research team or if you wish to talk with someone else. General information about participation in research studies can also be found at <a href="http://www.research.vcu.edu/human research/volunteers.htm">http://www.research.vcu.edu/human research/volunteers.htm</a>.

# CONSENT

I have been given the chance to read this consent form. I understand the information about this study. Questions that I wanted to ask about the study have been answered. My signature says that I am willing to participate in this study. I will receive a copy of the consent form once I have agreed to participate.

| Participant name printed | Participant signature | Da | Date |
|---|---|---|---|
| Name of Person Conducting Info | rmed Consent Discussion | | |
| Signature of Person Conducting I | nformed Consent Discussion | Date | |
| Principal Investigator Signature (i | f different from above) | Date | |